CLINICAL TRIAL: NCT03192696
Title: INSIGHT: EvaluatIoN of the PantheriS OCT- ImaGing AtHerectomy SysTem For Treatment of In-Stent Restenosis (ISR) Lesions In Lower Extremity Arteries
Brief Title: Pantheris Atherectomy Treatment of In-Stent Restenosis In Lower Extremity Arteries
Acronym: INSIGHT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Avinger, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P0942
Record Dates: First submitted 2017-06-12; First posted 2017-06-20 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Treatment Cohort (Experimental): Atherectomy of in-stent restenosis
  Interventions: Device: Atherectomy Catheter

INTERVENTIONS:
Device: Atherectomy Catheter — Treatment of restenotic lesions within stents previously placed within the artery.

SUMMARY:
A prospective, non-randomized, international, multi-center study to evaluate the safety and effectiveness of the Pantheris OCT-Imaging System to perform atherectomy in In-Stent Restenotic (ISR) lesions in lower extremity arteries.

DETAILED DESCRIPTION:
This is a prospective, global, single-arm, multi-center study to evaluate the safety and effectiveness of the Pantheris OCT-Imaging System to perform atherectomy of in-stent restenotic (ISR) lesions in lower extremity arteries.

The trial will enroll up to 140 subjects diagnosed with peripheral arterial disease of the lower extremities that have previously been treated with stenting at up to 20 sites. The primary disease must be located in reference vessel diameter of >3.0mm and ≤7.0mm. Trial success is focused on safety, including rates of major adverse events through 30 days as adjudicated by a Clinical Events Committee, and effectiveness, which will be evaluated using technical success defined as the percent of target lesions that have residual diameter stenosis <50% post-treatment with the Pantheris device alone as assessed by Angiographic Core Lab.

ELIGIBILITY:
Inclusion Criteria:

* Subject is >18 years old;
* Subject is willing and able to give informed consent;
* Subject has Rutherford Classification of I-V;
* Subject presenting with a single Class I, II or III ISR lesion as per Tosaka's Classification criteria in the lower leg extremities;
* Target lesion must be >70% stenosed and within a stented segment by angiographic visual estimation;
* Reference vessel lumen acceptable for treatment with Pantheris catheter size as per visual angiographic estimation;
* Target lesions must be within the stented segment and no more than 3 cm past the proximal or distal portions of the stent;
* Target lesion is ≤30 cm in length;
* Intraluminal crossing of totally occluded lesions prior to atherectomy;
* At least one patent tibial run-off vessel at baseline; and
* Subject is capable of meeting requirements and be present at the follow-up clinic visits at 30 days, 6 months and 12 months.

Exclusion Criteria:

* Subject is pregnant or breast feeding;
* Rutherford Class 0 or VI;
* Severe calcification of the target lesion;
* Acute ischemia and/or acute thrombosis of the target lesion segment;
* Target lesion with a covered stent;
* Target lesion in the iliac artery;
* Target lesion stenosis <70%;
* Target lesion >30 cm in length;
* Subjects with totally occluded stented segments that are not successfully crossed intraluminally prior to atherectomy treatment;
* Grade 4 or 5 stent fracture affecting target stent, or where evidence of stent protrusion into the lumen is noted on angiography in two orthogonal views;
* Subjects on chronic hemodialysis or creatinine level >2.5 mg/dL;
* CVA or stroke within 60 days prior to the index procedure;
* Endovascular or surgical procedure performed on the index limb less than or equal to 30 days prior to the index procedure;
* Planned endovascular or surgical procedure 30 days after the index procedure;
* Lesion in the contralateral limb requiring intervention during the index
* procedure or within 30 days of the index procedure;
* Known allergy to contrast agents or medications used to perform endovascular
* intervention that cannot be adequately pre-treated;
* Subjects in whom anti-platelet, aspirin, anticoagulant, or thrombolytic therapy is contraindicated;
* Any thrombolytic therapy within 2 weeks of the index procedure;
* Any clinical and/or angiographic complication attributed to the use of another device prior to the insertion of the study device into the subject during the index procedure;
* Subjects or their legal guardians who have not or will not sign the Informed Consent;
* Subjects who are unwilling or unable to comply with the follow-up study
* requirements; or
* Participation in any study of an investigational device, medication, biologic or other agent within 30 days prior to enrollment that is either a cardiovascular study or could, in the judgment of the investigator, affect the results of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2017-10-19 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Freedom from a composite of major adverse events (MAEs) through 30-day follow-up (safety) | Day 0 through 30 days post treatment procedure
  The primary safety endpoint is freedom from a composite of major adverse events (MAEs) through 30-day follow-up, as adjudicated by an independent CEC.
  Individual MAEs include:
  1. Cardiovascular-related death;
  2. Unplanned, major index limb amputation;
  3. Clinically driven target lesion revascularization (TLR);
  4. Myocardial infarction; or
  5. Device-associated events:
     1. Clinically significant perforation,
     2. Clinically significant dissection,
     3. Clinically significant embolus, or
     4. Pseudoaneurysm.
Technical success of Pantheris catheter treatment (efficacy) device | Day 0
  The primary efficacy endpoint of technical success is defined as the percent of target lesions that have a residual diameter stenosis <50% post the Pantheris device alone, as assessed by an independent Angiographic Core Laboratory.

SECONDARY OUTCOMES:
Stent structure freedom from new or worsening stent fracture post Pantheris treatment (safety) | Day 0
  Assess the stent for new or worsening stent fracture per comparative Pantheris OCT evaluation pre- and immediately post-procedure.
Secondary Effectiveness Endpoint - Freedom from TLR | 6 months post treatment procedure
  Freedom from TLR at 6 months as assessed by an independent CEC.
Secondary Effectiveness Endpoint - Procedural Success | Day 0
  Procedural success defined as the percent of target lesions that have residual diameter stenosis ≤ 30% post-Pantheris and any other adjunctive therapy, determined by independent Angiographic Core Laboratory.
Secondary Effectiveness Endpoint - Freedom from TLR | 12 months post treatment procedure
  Freedom from TLR at 12 months as assessed by an independent CEC.
Secondary Effectiveness Endpoint - Ankle-Brachial Index | 30 days, 6 and 12 months post treatment procedure
  Ankle-Brachial Index at 30 days, 6 and 12 months
Secondary Effectiveness Endpoint - Rutherford Classification | 30 days, 6 and 12 months post treatment procedure
  Rutherford Classification at 30 days, 6 and 12 months
Secondary Effectiveness Endpoint - Use Adjunctive Devices | Day 0
  Adjunctive devices (stent placement (bare metal or drug eluting stent), drug eluting balloon or other) utilized during the index procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Sean Janzer, MD, Principal Investigator — Einstein Medical Center
Locations (12):
- United States (12):
  - St. Bernards Medical Center, Jonesboro, Arkansas
  - Arkansas Heart Hospital, Little Rock, Arkansas
  - University of California San Diego (UCSD), San Diego, California
  - Advocate Christ Hospital and Medical Center, Oak Lawn, Illinois
  - Baton Rouge General Medical Center, Baton Rouge, Louisiana
  - University of Missouri, Columbia, Missouri
  - Deborah Heart and Lung Center, Browns Mills, New Jersey
  - TriHealth-Hatton Research Institute, Cincinnati, Ohio
  - Dayton Heart Center, Dayton, Ohio
  - Einstein Medical Center, Philadelphia, Pennsylvania
  - University of Tennessee Health Science Center, Memphis, Tennessee
  - Cardiovascular Associates of East Texas, Tyler, Texas

IPD SHARING:
Plan to Share IPD: No